CLINICAL TRIAL: NCT01524146
Title: To Establish a Multicenter Registry to Evaluate the Impact of Photodynamic Therapy in the Management of Patients With Unresectable Cholangiocarcinoma.
Brief Title: Photodynamic Therapy (PDT) Cholangiocarcinoma Registry
Acronym: PDTRegistry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1111012021
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Unresectable Cholangiocarcinoma; Biliary Obstruction; Stent Obstruction; Biliary Stricture
Keywords: Unresectable Cholangiocarcinoma; Biliary obstruction; Stent obstruction; Biliary stricture; Photodynamic therapy; PDT; Ablation
MeSH Terms: interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Photodynamic therapy: Subjects who will receive photodynamic therapy for palliation of unresectable Cholangiocarcinoma.
  Interventions: Procedure: Photodynamic Therapy

INTERVENTIONS:
Procedure: Photodynamic Therapy — PDT is a therapeutic approach that specifically targets neoplastic cells.
  • PDT involves three components:
  1. Photofrin or a similar Photosensitizing agent that would be injected 3 days prior to laser activation of the agent.
  2. Laser System - For laser energy delivery to activate the photosensitizing agent and induce tumor tissue necrosis
  3. Optic Fiber - Delivery Fiber used along with the laser system to achieve Photoactivation of the photosensitizing agent.
  Technique:
  Subjects will be injected with Photofrin or similar drug. 3 days post injection, the subject will receive photodynamic therapy during an Endoscopic Retrograde cholangiopancreatography (ERCP) procedure. Subject will undergo stenting as part of standard of care procedure post photodynamic therapy.
  Subject may undergo multiple photodynamic therapy sessions with a gap of at least 3 months.
  Other Names: PDT

SUMMARY:
Currently, very few centers offer Photodynamic therapy for unresectable Cholangiocarcinoma in the United States. Several European studies have reported the efficacy and safety of Photodynamic Therapy (PDT) for Cholangiocarcinoma, however, only a few studies have reported the same in the United States.

The establishment of a registry to capture all PDT cases within and outside US can help the investigators evaluate a larger and non-ambiguous sample population. This would help the investigators evaluate the technical success rates, clinical success rates, feasibility and safety of PDT for unresectable cholangiocarcinoma. With more endoscopists considering PDT as a therapeutic option along with adjuvant treatment for cholangiocarcinoma, there is a need to further evaluate the efficacy and safety of such combined procedures as well. The ultimate objective is to assess if PDT with or without additional or adjuvant treatment options prolongs survival duration and improves quality of life in patients with unresectable cholangiocarcinoma.

This multicenter registry has been initiated:

* To document the impact of PDT on the clinical management of unresectable cholangiocarcinoma.
* To assess the clinical and technical success rates of PDT for unresectable cholangiocarcinoma.

DETAILED DESCRIPTION:
PDT offers a number of practical advantages; it is minimally invasive and has a low complication rate, the procedure can easily be performed by a trained endoscopist, and it is well tolerated. In the trial conducted in Germany, the adverse events of PDT were mild to moderate, predictable, and relatively easy to control. Photosensitivity was the only systemic side effect (seen in only three patients). However, provided that simple guidelines for light exposure are followed, there is minimal risk to the patient, as shown by the low incidence of photosensitivity reactions in this study which all resolved.

A study from the Mayo group included 25 patients with unresectable cholangiocarcinoma who were treated with PDT from 1991 to 2004 showed that the time interval between diagnosis and treatment with PDT is an important predictor of survival following PDT even when adjusted for other potential factors that affect survival such as age, gender, Bismuth stage, presence of tumor mass on imaging and presence of extra biliary spread. Early treatment with PDT may lead to greater preservation of liver function. A recent study by the primary investigator has also recently reported improved survival in patients receiving PDT and stent compared to stent only (16.2 months vs 7.4 months).

Several other European studies have reported the efficacy and safety of PDT for cholangiocarcinoma; however, only a few studies have reported the same in the United States. This is again due to the fact that PDT is not offered as a therapeutic option for unresectable cholangiocarcinoma within US.

However, the establishment of a registry to capture all PDT cases within and outside US can help the investigators evaluate a larger and non ambiguous sample population. This would help the investigators evaluate the technical success rates, clinical success rates, feasibility and safety of PDT for unresectable cholangiocarcinoma.

The involvement of international sites is crucial, as the advanced endoscopists all over the world are offering photodynamic therapy for managing unresectable cholangiocarcinoma. However, because of the non-existence of a registry, and the fact that PDT is not offered in more than a few centers in the US; these cases are often reported with a smaller sample size. The registry hopes to combine all such comparable cases and collect enough relevant data for statistical analyses.

With more endoscopists considering PDT as a therapeutic option along with adjuvant treatment for cholangiocarcinoma, there is a need to further evaluate the efficacy and safety of such combined procedures as well. The ultimate objective is to assess if PDT with or without additional or adjuvant treatment options prolongs survival duration and improves quality of life in patients with unresectable cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is undergoing PDT for unresectable Cholangiocarcinoma
* Above 18 years of age

Exclusion Criteria:

* Any patient who will not undergo PDT for unresectable Cholangiocarcinoma
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from unresectable Cholangiocarcinoma who have a blocked bile duct or biliary stent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety | 3 years
  Documentation of Safety: Number of Participants with Adverse Events; Type, frequency and intensity of adverse events

SECONDARY OUTCOMES:
Efficacy | 3 years
  Documentation of efficacy: Technical and clinical success rates; and survival duration.
  Effectiveness will be assessed by visual inspection of tissue necrosis in the bile ducts one month post photo dynamic therapy delivery.
Concomitant Therapy Effect | 3 years
  Documentation of concomitant/adjuvant therapy and overall survival duration.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Weill Medical College of Cornell University, New York, New York

IPD SHARING:
Plan to Share IPD: No
No IPD Sharing